CLINICAL TRIAL: NCT03029390
Title: Effect of Administration of Berberine Versus Metformin on Glycemic Control, Insulin Sensitivity and Insulin Secretion in Patients With Prediabetes
Brief Title: Effect of Berberine Versus Metformin on Glycemic Control, Insulin Sensitivity and Insulin Secretion in Prediabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Karina Griselda Pérez Rubio, PhD, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BM-Prediabetes
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2022-06

CONDITIONS: Prediabetes; Impaired Fasting Glucose; Impaired Glucose Tolerance
Keywords: Prediabetes; hyperglycemia; Impaired Fasting Glucose; Metformin; Berberine; glucose intolerance
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Hyperglycemia | interventions — Berberine; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Berberine hydrochloride (Experimental): Berberine capsules, 500 mg, three per day before each meal during 12 weeks.
  The patients will have a forced titration period:
  First week they will receive one 500 mg capsule before breakfast Second week they will receive two 500 mg capsules (before breakfast and meal) From the third week until the end of the study, they will be receive three 500 mg capsules (before each meal)
  Interventions: Dietary Supplement: Berberine
- Metformin (Experimental): Metformin capsules, 850 mg, two per day before breakfast and dinner and one placebo capsule before lunch during 12 weeks.
  The patients will have a forced titration period:
  First week they will receive one 850 mg capsule before breakfast Second week they will receive one 500 mg capsules (before breakfast) and one placebo capsule (before meal).
  From the third week until the end of the study, they will be receive two 850 mg capsules (before breakfast and dinner) and one placebo capsule (before meal).
  Interventions: Drug: Metformin

INTERVENTIONS:
Dietary Supplement: Berberine — Berberine capsules, 500 mg, three per day before each meal during 14 weeks.
  The patients will have a running period during two weeks:
  First week they will receive one 500 mg capsule before breakfast Second week they will receive two 500 mg capsules (before breakfast and meal) From the third week until the end of the study (14 week), they will be receive three 500 mg
  Other Names: Berberine hydrochloride
  Arms: Berberine hydrochloride
Drug: Metformin — Metformin capsules, 850 mg, two per day before breakfast and dinner and one placebo capsule before lunch during 14 weeks.
  The patients will have a running period:
  First week they will receive one 850 mg capsule before breakfast Second week they will receive one 500 mg capsules (before breakfast) and one placebo capsule (before meal).
  From the third week until the end of the study (14 week), they will be receive two 850 mg capsules (before breakfast and dinner) and one placebo capsule (before meal).
  Arms: Metformin

SUMMARY:
Pre diabetes (PD) is a term that refers to alterations in glucose homeostasis, including impaired fasting glucose (IFG), Imparied glucose tolerance (IGT) or both, involving a higher risk to develop type 2 diabetes mellitus (T2DM) in 10 years.

The efficacy of pharmacotherapy in the prevention of diabetes in adults with prediabetes has been demonstrated, the first line of pharmacology treatment is metformin, on the other hand, the traditional Chinese and Ayurverica medicine offer potential active substances for the treatment of hyperglucemia like berberine.

Berberine is an extract with hypoglycemic effects in animal models as well as in clinical trials in type 2 diabetes mellitus even compared to metformin, for this reason comparing it's activity against metformin in prediabetes would provide impact information on a new alternative treatment and compare with the standard pharmacological treatment.

The aim of the study evaluate the effect of administration of berberine versus metaformine on glycemic control, insulin secretion and insulin sensitivity in patients with pre diabetes.

The investigators hypothesis is that the administration of berberine versus metformin modifies glycemic control, insulin sensitivity and insulin secretion in patients with prediabetes.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial in 28 patients with a diagnosis of prediabetes (IFG and IGT) in accordance with the American Diabetes Association with out treatment.

They will be assigned randomly two groups of 14 patients, one of the groups will receive 850 mg of metformin twice at day (before breakfast and before dinner) and one pill of placebo (before lunch) for 14 weeks. There will be a running period, starting with a dose of 500 mg the first week, the second week increasing to 1000 mg and from the third to the fourteenth week will be a dose of 1500 mg.

The other group will receive 500 mg of berberine three times at day (each one before the mealtime) for14 weeks. There will be a running period, starting with a dose of 850 mg the first week, the second week dose of 850 mg of metformin plus one placebo pill and from the third week to the fourteenth week will be a dose of 1700 mg ( two 850 mg metformin pills) plus one placebo pill.

They will be measured fasting blood glucose, postprandial glucose levels and glycosylated hemoglobin, and will be calculated Area Under Curve of glucose and insulin, total insulin secretion (Insolinogenic index), first-phase of insulin secretion (Strumvoll index) and insulin sensitivity (Matsuda index).

This protocol it's already approved by the local ethics committee and written informed consent it's going to be obtained from all volunteers.

Statistical analysis will be presented through measures of central tendency and dispersion, average and deviation standard for quantitative variables; frequencies and percentage for qualitative variable. Qualitative variables will be analyzed by X2, will be used for differences inter-group Mann-Whitney U Test and Wilcoxon Test for the within-groups differences. It will be considered statistical significance p≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients both sexes
* Age between 31 and 60 years
* Diagnosis of prediabetes according 2 ADA criteria (fasting blood glucose levels between 100-125 mg/dl and postprandial blood glucose levels after an oral glucose tolerance test with 75 of oral glucose between 140-199 mg/dl)
* Body Mass Index from 25 to 34.9kg/m2
* Informed consent signed

Exclusion Criteria:

* Women with confirmed or suspected pregnancy
* Women under lactation and/or puerperium
* Hypersensibility to ingredients of intervention
* Physical impossibility for taking pills
* Known uncontrolled renal, hepatic, heart or thyroid diseased
* Diabetes diagnosis
* Previous treatment for glucose
* Body Mass Index ≥35 kg/m2
* Glycosylated hemoglobin > 6.5%
* Triglycerides ≥500 mg/dL
* Total cholesterol ≥240 mg/dL
* Low density lipoprotein (c-LDL) ≥190 mg/dL
* Blood Pressure ≥140/90 mmHg

Ages: 31 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-02 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Fasting glucose levels | Baseline to week 14
  The fasting glucose levels will be evaluated at baseline and week 14 with enzymatic/ colorimetric techniques and the entered values reflect the fasting glucose level at week 14
postprandial glucose levels | baseline to week 14
  Postprandial glucose will be evaluated at baseline week 14 after a oral glucose tolerance test with enzymatic/ colorimetric techniques and the entered values reflect the insulin sensitivity at week 14
Glycosylated hemoglobin | baseline to week 14
  Glycosylated hemoglobin will be evaluated at baseline and week 14 by Elisa and the entered values reflect the glycosylated hemoglobin at week 14
Total insulin secretion | baseline to week 14
  Total insulin secretion will be calculated at baseline and week 14 with insulinogenic index and the entered values reflect the total insulin secretion at week 14
First phase of insulin secretion | baseline to week 14
  The first phase of insulin secretion will be calculated at baseline and week 14 with Strumvoll index and the entered values reflect the first phase of insulin secretion at week 14
Insulin sensitivity | baseline to week 14
  Insulin sensitivity will be calculated at baseline and week 14 with Matsuda index and the entered values reflect the insulin sensitivity at week 14

SECONDARY OUTCOMES:
Body Weight | Baseline to week 14
  The body weight will be measured at baseline, week 3, week 6, week 10, and week 14 with a bioimpedance balance and the entered values reflect the body weight at week 14
Body Mass Index | Baseline to week 14
  Body Mas Index will be calculated at baseline, week 3, week 6, week 10, and week 14 with the Quetelet index formula and the entered values reflect the body mass index at week 14
Body fat percentage | Baseline to week 14
  Body fat percentage will be evaluated at baseline, week 3, week 6, week 10, and week 14 by Bioimpedance technique and the entered values reflect the body fat percentage at week 14
Waist circumference | Baseline to week 14
  Waist circumference will be evaluated at baseline, week 3, week 6, week 10 and week 14 by World Health Organization technique and the entered values reflect the waist circumference mesure at week 14
Blood pressure | Baseline to week 14
  Blood pressure will be measured at baseline,week 3, week 6, week 10 and week week 14 with a digital sphygmomanometer and the entered values reflect the blood pressure at week 14
Total cholesterol | Baseline to week 14
  Total cholesterol levels will be evaluated at baseline and week 14 by enzymatic/colorimetric techniques and the entered values reflect the total cholesterol level at week 14
Triglycerides levels | Baseline to week 14
  Triglycerides levels will be evaluated at baseline and week 14 with enzymatic/colorimetric techniques and the entered values reflect the triglycerides level at week 14
High density lipoprotein (c-HDL) levels | Baseline to week 14
  c-HDL levels will be evaluated at baseline and week 14 with enzymatic/colorimetric techniques and the entered values reflect the c-HDL level at week 14
Low density lipoprotein (c-LDL) levels | Baseline to week 14
  c-LDL levels will be will be calculated at baseline and week 14 with Friedewald Formula and the entered values reflect the c-HDL level at week 14
Alanine aminotransferase (ALT) levels | Baseline to week 14
  ALT levels will be evaluated at baseline and week 14 with enzymatic/colorimetric techniques
Aspartate aminotransferase (AST) levels | Baseline to week 14
  AST levels will be evaluated at baseline and week 14 with enzymatic/colorimetric techniques
Creatinine levels | Baseline to week 14
  Creatinine levels will be evaluated at baseline and week 14 with enzymatic/colorimetric techniques

CONTACTS AND LOCATIONS:
Overall Officials: KARINA GRISELDA PEREZ, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Instituto de Terapeútica Experimental y Clínica. Centro Universitario de Ciencias de la Salud. Universidad de Guadalajara, Guadalajara, Jalisco, Mexico